CLINICAL TRIAL: NCT02079753
Title: Oxygenation Using a Single Portable Pulse-dose-conserving Device Compared to Combined Use of Stationary and Portable Oxygen Delivery Devices.
Brief Title: Single Portable Pulse-dose-conserving Device vs. Combined Use of Stationary and Portable.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Son Espases (Other)
Collaborators: Linde AG (Industry)
Responsible Party: Principal Investigator, Aina M Yañez, Epidemilogist, Hospital Son Espases
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: POCs
Record Dates: First submitted 2014-02-27; First posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD, portable concentrator, oxygen sources
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combined system (Active Comparator): During the first visit, the technician installed a reservoir of liquid oxygen (Liberator 30, Caire) and a liquid Stroller oxygen pack (Caire) for patients using liquid oxygen, or a VisionAire5 (Airsep) stationary concentrator and an Inogen One G2 portable (Inogen) concentrator for patients using concentrators.
  Interventions: Device: Combination system of a portable and a stationary device.
- single system (Experimental): Inogen One G2 portable concentrator (Inogen)
  Interventions: Device: Inogen

INTERVENTIONS:
Device: Inogen — single pulse dose concentrator (Inogen One G2 portable. Inogen) device for 24 hours
  Arms: single system
Device: Combination system of a portable and a stationary device. — Combination system of a portable and a stationary device (reservoir of liquid oxygen "Liberator 30, Caire" and a liquid Stroller oxygen pack "Caire" for patients using previously liquid oxygen, or a VisionAire5 "Airsep" stationary concentrator and an Inogen One G2 portable "Inogen" concentrator for patients using previously concentrators)
  Arms: combined system

SUMMARY:
Introduction: Portable oxygen devices simplify and facilitate patient therapy. This study was designed to compare oxygen saturation and patient satisfaction with a portable oxygen concentrator or with a combined system consisting of a fixed device with continuous flow oxygen dispensation and a portable device with pulse dispensation for ambulation.

Methods: This cross-over trial assessed 25 patients with COPD (92% men; mean age 72.2 ± 7.4 years; mean FEV 34.14 ± 12.51%) at four hospitals in Madrid. All patients had previously used the combined system, consisting of a fixed oxygenation system and a portable system for ambulation, with 16 (64%) using stationary and portable concentrators and 9 (36%) using a stationary reservoir and portable liquid oxygen bag. Oxygenation settings at rest and while walking were determined at baseline. Patients were maintained on the previous combined system for one week and then switched to the portable oxygen concentrator for one week. Mean SpO2 over 24 hours was calculated by the software in the oximeter, and compliance was monitored

ELIGIBILITY:
Inclusion Criteria:

* aged 40-80 years
* had been diagnosed with COPD following the GOLD criteria
* were receiving oxygen therapy using a fixed oxygenation system and a portable system for ambulation
* without exacerbation during the previous month
* agreed to participate

Exclusion Criteria:

* terminally ill
* unable to understand Spanish
* had high oxygen flow at rest (> 3 lpm)
* high respiratory frequency at rest (> 32 rpm)
* were not achieving adequate O2 saturation levels during titration with the portable oxygen source
* had previously been diagnosed with obstructive sleep apnea hypopnea syndrome (SAHS)
* were receiving mechanical ventilation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Percentage of time desaturated below 90% when using a combined oxygenation system | at day 7
  oxygenation of patient during use of a combined system consisting of a fixed device with continuous flow oxygen dispensation and a portable device with pulse dispensation for ambulation.
Percentage of time desaturated below 90% using single oxygenation system | day 14
  Oxygenation of patient during use of a portable oxygen pulse dose concentrator.

CONTACTS AND LOCATIONS:
Locations (1):
- Servicio de Neumología. Hospital Clínico de San Carlos. Facultad de medicina. Universidad complutense de Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Yanez AM, Prat JP, Alvarez-Sala JL, Calle M, Diaz Lobato S, Garcia Gonzalez JL, Rodriguez Gonzalez-Moro JM, Galera-Martinez R, Villasante C, Ramos I, Franco-Gay M, de Lucas P. Oxygenation With a Single Portable Pulse-Dose Oxygen-Conserving Device and Combined Stationary and Portable Oxygen Delivery Devices in Subjects With COPD. Respir Care. 2015 Mar;60(3):382-7. doi: 10.4187/respcare.03470. Epub 2014 Nov 25. PMID 25425710